CLINICAL TRIAL: NCT04803019
Title: Transarterial Embolization Alone Versus Drug-Eluting Beads Chemoembolization for Hepatocellular Carcinoma. A Randomized Controlled Trial
Brief Title: Transarterial Embolization Alone Versus Drug-Eluting Beads Chemoembolization for Hepatocellular Carcinoma
Acronym: RAD-18-TAcE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Rita Golfieri, Professor, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAD-18-TAcE
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Microspheres; Embolization, Therapeutic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEB-TACE or chemoembolization with microspheres (Active Comparator): The chemotherapy used in this arm is the Doxorubicin that will be carried into the tumor by Embozene TANDEM® (Boston Scientific) microspheres. TANDEM® embozene microspheres are made of non-resorbable, biocompatible, hydrogel microspheres, subjected to precision calibration and coated with an inorganic perfluorate polymer (Polyzene®-F)
  Interventions: Combination Product: DEB-TACE
- TAE or embolization with microspheres (Active Comparator): The TAE will be performed with Embozene microspheres (Boston Scientific). Embozene microspheres are spherical particles of hydrogel, precisely calibrated, biocompatible, non-absorbable and coated with a perfluorinated inorganic polymer (Polyzene®-F)
  Interventions: Device: TAE

INTERVENTIONS:
Combination Product: DEB-TACE — The chemotherapy used in this arm is the Doxorubicin that will be carried into the tumor by Embozene TANDEM® (Boston Scientific) microspheres. TANDEM® embozene microspheres are made of non-resorbable, biocompatible, hydrogel microspheres, subjected to precision calibration and coated with an inorganic perfluorate polymer (Polyzene®-F).
  TANDEM® embozene microspheres are available in three different sizes, in 2 ml and 3 ml volumes of product and are supplied in preloaded vials and syringes.The maximum loadable amount on the hydrospheres 50 mg of Doxorubicina for ml. The maximum injectable dose of Doxorubicin for each treatment is 150 mg and therefore the maximum amount of microspheres that can be used for each treatment is 3 ml. The size of microspheres that will be used in this study is up to 100 ± 25 μm.
  Other Names: Chemoembolization with microspheres
  Arms: DEB-TACE or chemoembolization with microspheres
Device: TAE — The TAE will be performed with Embozene microspheres (Boston Scientific). Embozene microspheres are spherical particles of hydrogel, precisely calibrated, biocompatible, non-absorbable and coated with a perfluorinated inorganic polymer (Polyzene®-F). This medical device is available in various sizes; in this study, to avoid that the particle size exceeds the one used for the treatment of arm A, it will be possible to use microspheres with dimensions up to 100 μm (range 75 ± 125 μm).
  Embozene microspheres are offered in vials containing 1 ml of suspended product in physiological saline solution for apyrogenic sterile transport. The total volume of the Embozene microspheres, including the transport solution, is about 7 ml. To this product it is necessary to add an appropriate amount of non-ionic contrast medium in order to obtain a homogeneous suspension and with good visibility during the injection under fluoroscopy.
  Other Names: Embolization with microspheres
  Arms: TAE or embolization with microspheres

SUMMARY:
Developed in Japan in the 1980s, TACE became the most frequent treatment for unresectable hepatocellular carcinoma (HCC) in patients with preserved hepatic function after 2002, when two radiochemotherapies (RCTs) showed survival benefits for HCC patients who underwent conventional Lipiodol-based TACE (cTACE). Nowadays, nearly half of HCC patients undergo this procedure during their clinical history. In the last ten years, cTACE has been challenged by an alternative procedure, drug-eluting beads-TACE (DEB-TACE), after the introduction of calibrated embolizing microspheres loaded with a chemotherapeutic agent. DEB-TACE is considered to be less toxic and better standardized than cTACE, with reported no differences in patient survival. Since 2006, DEB-TACE has become the standard in many centers worldwide. Though, the need of adding doxorubicin to small beads embolization alone (TAE) remains unsettled. Though cTACE/DEB-TACE and TAE have been compared in several RCTs, no study demonstrated a clear survival benefit associated with the former.

Our study aims to compare first-line DEB-TACE and TAE on a random sample of HCC with the hypothesis that the addition of drug to embolization with small size beads is not associated with a survival benefit when compared to embolization alone performed with tiny calibrated microspheres. HCC is considered a chemo-resistant tumor and to date there is no clear evidence of benefits in associating anticancer agents to TAE. On the other hand, the optimal size of embolic agents has still to be defined. A comparative evaluation of TACE and TAE is essential for two additional reasons: a) it is still unclear whether side effects following embolization procedures are related to the embolization itself, to drug addition or both; b) DEB-TACE procedure is more expensive than TAE and, given the current attention on cancer-related health care cost control, identification of opportunities for cost savings in HCC treatments of an increasingly common cancer would be valuable.

DETAILED DESCRIPTION:
Specific Aims

Specific aim 1 Compare time to progression (TTP) treated with TAE and DEB-TACE in a homogeneous hepatocellular carcinoma (HCC) patient population

Specific aim 2 Compare

* safety - severe adverse events (SAE)
* radiologic tumor response (mRECIST)
* overall survival (OS)
* cost-effectiveness after the entire follow-up

Study plan

Experimental design This is an interventional with drug, multicenter, prospective, randomized open label study.

Experimental design Aim 1 The study was designed, in relation to the primary endpoint, as an equivalence trial between two intra-arterial HCC treatments, i.e. DEB-TACE and TAE. The TTP considered as the reference value for the DEB-TACE arm is 9 months, on the basis of the results of our previous multicentric experience. The study is designed as an equivalence trial on the primary endpoint. The standard deviation of TTP is expected not to exceed 6 months, through accurate selection criteria of included patients. The equivalence limit is set to no more than 5 months between the two arms. Thus, using appropriate formulae each arm will be formed by 69 patients (alpha:0.05; beta:0.80). Taking into account a 10% of drop-out, the final sample size per each arm will be of 77 patients (154 total).

Experimental design Aim 2

* Safety. Adverse events (AEs) and severe adverse events (SAEs) will be monitored and recorded. AE will be assessed during and after each treatment and at all follow-up visits and graded according to the NCI Common Terminology Criteria for AE (CTCAE) version 3.0. The AEs occurring within 4 weeks after TACE will be considered as treatment related. SAE incidence in both arms will be ascertained assuming a reduction of SAE from 25% after TACE to 19% after TAE (25% of reduction). Such an assumption would require 607 patients per arm for being confirmed. To accomplish this task, the O'Brien-Fleming stopping boundaries will be applied considering an analysis when 69 patients for each arm will be obtained and follow-up ended. Applying stopping boundaries to this sample size, a nominal p-value <0.001 (z-score: 3.15) is needed to confirm the assumption. If the p-value will be above this threshold (even if <0.05) the null hypothesis will be not refused.
* Efficacy. The response will be evaluated by CT or MRI as local (per-lesion) response and overall (per-patient) response, according to mRECIST, at 1 month after each TACE and, thereafter, every 3 months, for at least 2 years.
* Survival. Through the selection previously described, we expected a standard deviation of the mean survival of no more than 10 months. To design the present equivalence trial we also expected a difference in the mean survival not greater than 5 months (equivalence limit) between the two groups. Using formulas proposed by Julious et al., each arm will be formed by 69 patients (alpha: 0.05; beta: 0.80). To obtain more robust estimate and accounting for possible dropout from the study a 10% of patients will be added to the initial sample size, resulting in 77 patients for each arm.
* Cost-effectiveness will be assessed from a third payer perspective, thus, including only direct costs of the procedures and related costs (hospitalization, imaging, etc.). The effectiveness will be assessed by measuring the life-expectancy. Incremental cost-effectiveness ratio (ICER) will be used to evaluate the cost-effectiveness of one treatment over the counterpart.

Study population The study involves the enrollment of a total of 154 patients, 77 per randomization arm, with a HCC diagnosis, according to the guidelines of the American Association for the Study of the Liver Disease (AASLD), as in clinical practice. The enrolled patients will have to meet the inclusion criteria and sign the informed consent for the participation in this study. At the time of enrollment, demographic, clinical and radiological data will be collected, as in standard clinical practice.

Treatment

Treatment study In the present study, only patients in the DEB-TACE arm (Arm A) will receive intra-arterial hepatic chemotherapy (Doxorubicin). Both treatment arms, on the other hand, will receive arterial embolization of the branches that vascularize the tumor lesions.

Arm A: DEB-TACE or chemoembolization with microspheres. The chemotherapy used in this arm is the Doxorubicin that will be carried into the tumor by Embozene TANDEM® (Boston Scientific) microspheres. TANDEM® embozene microspheres are made of non-resorbable, biocompatible, hydrogel microspheres, subjected to precision calibration and coated with an inorganic perfluorate polymer (Polyzene®-F). Thanks to their design, the microspheres can be loaded with drugs, such as doxorubicin, in order to administer a local, controlled and constant dose of the drug to the tumor sites affected after embolization.

TANDEM® embozene microspheres are available in three different sizes, in 2 ml and 3 ml volumes of product and are supplied in preloaded vials and syringes.The maximum loadable amount on the hydrospheres 50 mg of Doxorubicina for ml. The maximum injectable dose of Doxorubicin for each treatment is 150 mg and therefore the maximum amount of microspheres that can be used for each treatment is 3 ml. The size of microspheres that will be used in this study is up to 100 ± 25 μm.

Arm B: TAE or embolization with microspheres. The TAE will be performed with Embozene microspheres (Boston Scientific). Embozene microspheres are spherical particles of hydrogel, precisely calibrated, biocompatible, non-absorbable and coated with a perfluorinated inorganic polymer (Polyzene-F). This medical device is available in various sizes; in this study, to avoid that the particle size exceeds the one used for the treatment of arm A, it will be possible to use microspheres with dimensions up to 100 μm (range 75 ± 125 μm).

Embozene microspheres are offered in vials containing 1 ml of suspended product in physiological saline solution for apyrogenic sterile transport. The total volume of the Embozene microspheres, including the transport solution, is about 7 ml. To this product it is necessary to add an appropriate amount of non-ionic contrast medium in order to obtain a homogeneous suspension and with good visibility during the injection under fluoroscopy.

In enrolled patients, regardless of the treatment arm, the possible presence of extra-hepatic shunts, such as gastric and pulmonary arteries arising from the hepatic branches, should be appropriately assessed. As in standard radiological practice in case of intra-arterial hepatic treatments, if these shunts are macroscopically evident, the preventive closure of the same vessels will be evaluated, using the devices that will be more suitable on a case-by-case basis. If these shunts are not treatable by occlusive devices, the enrolled patient will not be treated in the clinical study and the patient will be considered as drop-out. Both treatments will be repeated "on demand" after demonstration to the imaging of the presence of vital tumor ie absence of complete response (complete response, CR) or in case of intrahepatic distal recurrence at follow-up.

Safety assessment The evaluation of the safety of the experimental treatment will consist in the monitoring and recording of AEs and SAEs.

ELIGIBILITY:
Inclusion Criteria:

- First level eligibility criteria include

1. HCC diagnosis according to the AASLD criteria [26];
2. patients ≥18 years;
3. HCC unsuitable for curative treatment or had failed/recurred after resection/ablation diagnosed according to the AASLD criteria;
4. no previous treatment in target lesions (prior treatments including resection on non-target lesions will be accepted);
5. Child-Pugh class A or B (max score 7);
6. ECOG Performance Status (PS) <2;
7. target lesion measurable according to mRECIST.

Second level eligibility criteria include:

1. The modified hepatoma arterial-embolization prognostic score (m-HAP-II), based on bilirubin, albumin, serum alpha fetoprotein, tumor number and tumor size, divides patients in 4 classes (A, B, C, D) with different survivals and is useful for prognosis stratification. The first selection criteria will be m-HAP-II classes B or C fulfilment.
2. The UNOS/TNM stage: only patients with T1, T2, T3 and T4 tumors will be included.

   These two main criteria will be used for stratification of patients prior to randomization in order to obtain identical prevalence of m-HAP-II classes B/C and of UNOS/TNM stages from T1 to T4a
3. obtaining of the informed consent.

Exclusion Criteria:

1. infiltrative HCC;
2. neoplastic branch or main portal vein invasion;
3. equivocal hepatic lesion;
4. advanced liver disease (bilirubin levels >2.5 mg dl-1, albumin <30 g l-1, platelets <50 x 109/L, INR >1.5);
5. ascites and/or F3 oesophageal varices;
6. other tumors in the previous 5 years;
7. technical contraindications to arteriography or TACE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2019-12-04 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Time to progression | The TTP considered as the reference value is 9 months
  TTP since randomization, as recommended from expert panel opinion, after TAE and DEB-TACE

CONTACTS AND LOCATIONS:
Overall Officials: Rita Golfieri, Professor, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Llovet JM, Real MI, Montana X, Planas R, Coll S, Aponte J, Ayuso C, Sala M, Muchart J, Sola R, Rodes J, Bruix J; Barcelona Liver Cancer Group. Arterial embolisation or chemoembolisation versus symptomatic treatment in patients with unresectable hepatocellular carcinoma: a randomised controlled trial. Lancet. 2002 May 18;359(9319):1734-9. doi: 10.1016/S0140-6736(02)08649-X. PMID 12049862
- [Background] Lo CM, Ngan H, Tso WK, Liu CL, Lam CM, Poon RT, Fan ST, Wong J. Randomized controlled trial of transarterial lipiodol chemoembolization for unresectable hepatocellular carcinoma. Hepatology. 2002 May;35(5):1164-71. doi: 10.1053/jhep.2002.33156. PMID 11981766
- [Background] Geschwind JF, Kudo M, Marrero JA, Venook AP, Chen XP, Bronowicki JP, Dagher L, Furuse J, Ladron de Guevara L, Papandreou C, Sanyal AJ, Takayama T, Ye SL, Yoon SK, Nakajima K, Lehr R, Heldner S, Lencioni R. TACE Treatment in Patients with Sorafenib-treated Unresectable Hepatocellular Carcinoma in Clinical Practice: Final Analysis of GIDEON. Radiology. 2016 May;279(2):630-40. doi: 10.1148/radiol.2015150667. Epub 2016 Jan 8. PMID 26744927
- [Background] Park JW, Chen M, Colombo M, Roberts LR, Schwartz M, Chen PJ, Kudo M, Johnson P, Wagner S, Orsini LS, Sherman M. Global patterns of hepatocellular carcinoma management from diagnosis to death: the BRIDGE Study. Liver Int. 2015 Sep;35(9):2155-66. doi: 10.1111/liv.12818. Epub 2015 Mar 25. PMID 25752327
- [Background] Golfieri R, Giampalma E, Renzulli M, Cioni R, Bargellini I, Bartolozzi C, Breatta AD, Gandini G, Nani R, Gasparini D, Cucchetti A, Bolondi L, Trevisani F; PRECISION ITALIA STUDY GROUP. Randomised controlled trial of doxorubicin-eluting beads vs conventional chemoembolisation for hepatocellular carcinoma. Br J Cancer. 2014 Jul 15;111(2):255-64. doi: 10.1038/bjc.2014.199. Epub 2014 Jun 17. PMID 24937669
- [Background] Sergio A, Cristofori C, Cardin R, Pivetta G, Ragazzi R, Baldan A, Girardi L, Cillo U, Burra P, Giacomin A, Farinati F. Transcatheter arterial chemoembolization (TACE) in hepatocellular carcinoma (HCC): the role of angiogenesis and invasiveness. Am J Gastroenterol. 2008 Apr;103(4):914-21. doi: 10.1111/j.1572-0241.2007.01712.x. Epub 2008 Jan 2. PMID 18177453
- [Background] Shim JH, Park JW, Kim JH, An M, Kong SY, Nam BH, Choi JI, Kim HB, Lee WJ, Kim CM. Association between increment of serum VEGF level and prognosis after transcatheter arterial chemoembolization in hepatocellular carcinoma patients. Cancer Sci. 2008 Oct;99(10):2037-44. doi: 10.1111/j.1349-7006.2008.00909.x. PMID 19016764
- [Background] Brown KS. Chemotherapy and other systemic therapies for hepatocellular carcinoma and liver metastases. Semin Intervent Radiol. 2006 Mar;23(1):99-108. doi: 10.1055/s-2006-939845. PMID 21326724
- [Background] Varela M, Real MI, Burrel M, Forner A, Sala M, Brunet M, Ayuso C, Castells L, Montana X, Llovet JM, Bruix J. Chemoembolization of hepatocellular carcinoma with drug eluting beads: efficacy and doxorubicin pharmacokinetics. J Hepatol. 2007 Mar;46(3):474-81. doi: 10.1016/j.jhep.2006.10.020. Epub 2006 Nov 29. PMID 17239480
- [Background] Marelli L, Stigliano R, Triantos C, Senzolo M, Cholongitas E, Davies N, Tibballs J, Meyer T, Patch DW, Burroughs AK. Transarterial therapy for hepatocellular carcinoma: which technique is more effective? A systematic review of cohort and randomized studies. Cardiovasc Intervent Radiol. 2007 Jan-Feb;30(1):6-25. doi: 10.1007/s00270-006-0062-3. PMID 17103105
- [Background] Tsochatzis EA, Meyer T, Burroughs AK. Hepatocellular carcinoma. N Engl J Med. 2012 Jan 5;366(1):92; author reply 92-3. doi: 10.1056/NEJMc1112501. No abstract available. PMID 22216857
- [Background] Poon RT, Tso WK, Pang RW, Ng KK, Woo R, Tai KS, Fan ST. A phase I/II trial of chemoembolization for hepatocellular carcinoma using a novel intra-arterial drug-eluting bead. Clin Gastroenterol Hepatol. 2007 Sep;5(9):1100-8. doi: 10.1016/j.cgh.2007.04.021. Epub 2007 Jul 12. PMID 17627902
- [Background] Cucchetti A, Trevisani F, Cappelli A, Mosconi C, Renzulli M, Pinna AD, Golfieri R. Cost-effectiveness of doxorubicin-eluting beads versus conventional trans-arterial chemo-embolization for hepatocellular carcinoma. Dig Liver Dis. 2016 Jul;48(7):798-805. doi: 10.1016/j.dld.2016.03.031. Epub 2016 May 20. PMID 27263056
- [Background] Malagari K, Pomoni M, Kelekis A, Pomoni A, Dourakis S, Spyridopoulos T, Moschouris H, Emmanouil E, Rizos S, Kelekis D. Prospective randomized comparison of chemoembolization with doxorubicin-eluting beads and bland embolization with BeadBlock for hepatocellular carcinoma. Cardiovasc Intervent Radiol. 2010 Jun;33(3):541-51. doi: 10.1007/s00270-009-9750-0. Epub 2009 Nov 24. PMID 19937027
- [Background] Meyer T, Kirkwood A, Roughton M, Beare S, Tsochatzis E, Yu D, Davies N, Williams E, Pereira SP, Hochhauser D, Mayer A, Gillmore R, O'Beirne J, Patch D, Burroughs AK. A randomised phase II/III trial of 3-weekly cisplatin-based sequential transarterial chemoembolisation vs embolisation alone for hepatocellular carcinoma. Br J Cancer. 2013 Apr 2;108(6):1252-9. doi: 10.1038/bjc.2013.85. Epub 2013 Feb 28. PMID 23449352
- [Background] Brown KT, Do RK, Gonen M, Covey AM, Getrajdman GI, Sofocleous CT, Jarnagin WR, D'Angelica MI, Allen PJ, Erinjeri JP, Brody LA, O'Neill GP, Johnson KN, Garcia AR, Beattie C, Zhao B, Solomon SB, Schwartz LH, DeMatteo R, Abou-Alfa GK. Randomized Trial of Hepatic Artery Embolization for Hepatocellular Carcinoma Using Doxorubicin-Eluting Microspheres Compared With Embolization With Microspheres Alone. J Clin Oncol. 2016 Jun 10;34(17):2046-53. doi: 10.1200/JCO.2015.64.0821. Epub 2016 Feb 1. PMID 26834067
- [Background] Massarweh NN, Davila JA, El-Serag HB, Duan Z, Temple S, May S, Sada YH, Anaya DA. Transarterial bland versus chemoembolization for hepatocellular carcinoma: rethinking a gold standard. J Surg Res. 2016 Feb;200(2):552-9. doi: 10.1016/j.jss.2015.09.034. Epub 2015 Oct 3. PMID 26507276
- [Background] Osuga K, Hori S, Hiraishi K, Sugiura T, Hata Y, Higashihara H, Maeda N, Tomoda K, Nakamura H. Bland embolization of hepatocellular carcinoma using superabsorbent polymer microspheres. Cardiovasc Intervent Radiol. 2008 Nov-Dec;31(6):1108-16. doi: 10.1007/s00270-008-9369-6. Epub 2008 Jun 10. PMID 18543028
- [Background] Takayasu K, Arii S, Ikai I, Omata M, Okita K, Ichida T, Matsuyama Y, Nakanuma Y, Kojiro M, Makuuchi M, Yamaoka Y; Liver Cancer Study Group of Japan. Prospective cohort study of transarterial chemoembolization for unresectable hepatocellular carcinoma in 8510 patients. Gastroenterology. 2006 Aug;131(2):461-9. doi: 10.1053/j.gastro.2006.05.021. PMID 16890600
- [Background] Tsochatzis E, Meyer T, Marelli L, Burroughs AK. Which transarterial therapy is best for hepatocellular carcinoma?--the evidence to date. J Hepatol. 2010 Sep;53(3):588. doi: 10.1016/j.jhep.2010.01.031. Epub 2010 Mar 24. No abstract available. PMID 20472319
- [Background] Tsochatzis E, Meyer T, O'Beirne J, Burroughs AK. Transarterial chemoembolisation is not superior to embolisation alone: the recent European Association for the Study of the Liver (EASL) - European Organisation for Research and Treatment of Cancer (EORTC) guidelines. Eur J Cancer. 2013 Apr;49(6):1509-10. doi: 10.1016/j.ejca.2012.11.012. Epub 2012 Dec 8. No abstract available. PMID 23231982
- [Background] Llovet JM, Di Bisceglie AM, Bruix J, Kramer BS, Lencioni R, Zhu AX, Sherman M, Schwartz M, Lotze M, Talwalkar J, Gores GJ; Panel of Experts in HCC-Design Clinical Trials. Design and endpoints of clinical trials in hepatocellular carcinoma. J Natl Cancer Inst. 2008 May 21;100(10):698-711. doi: 10.1093/jnci/djn134. Epub 2008 May 13. PMID 18477802
- [Background] Lencioni R, Llovet JM. Modified RECIST (mRECIST) assessment for hepatocellular carcinoma. Semin Liver Dis. 2010 Feb;30(1):52-60. doi: 10.1055/s-0030-1247132. Epub 2010 Feb 19. PMID 20175033
- [Background] Julious SA. Sample sizes for clinical trials with normal data. Stat Med. 2004 Jun 30;23(12):1921-86. doi: 10.1002/sim.1783. PMID 15195324
- [Background] Bruix J, Reig M, Sherman M. Evidence-Based Diagnosis, Staging, and Treatment of Patients With Hepatocellular Carcinoma. Gastroenterology. 2016 Apr;150(4):835-53. doi: 10.1053/j.gastro.2015.12.041. Epub 2016 Jan 12. PMID 26795574
- [Background] Park Y, Kim SU, Kim BK, Park JY, Kim DY, Ahn SH, Park YE, Park JH, Lee YI, Yun HR, Han KH. Addition of tumor multiplicity improves the prognostic performance of the hepatoma arterial-embolization prognostic score. Liver Int. 2016 Jan;36(1):100-7. doi: 10.1111/liv.12878. Epub 2015 Jun 22. PMID 26013186
- [Background] Cappelli A, Cucchetti A, Cabibbo G, Mosconi C, Maida M, Attardo S, Pettinari I, Pinna AD, Golfieri R. Refining prognosis after trans-arterial chemo-embolization for hepatocellular carcinoma. Liver Int. 2016 May;36(5):729-36. doi: 10.1111/liv.13029. Epub 2015 Dec 23. PMID 26604044
- [Background] Italian Association for the Study of the Liver (AISF); AISF Expert Panel; AISF Coordinating Committee; Bolondi L, Cillo U, Colombo M, Craxi A, Farinati F, Giannini EG, Golfieri R, Levrero M, Pinna AD, Piscaglia F, Raimondo G, Trevisani F, Bruno R, Caraceni P, Ciancio A, Coco B, Fraquelli M, Rendina M, Squadrito G, Toniutto P. Position paper of the Italian Association for the Study of the Liver (AISF): the multidisciplinary clinical approach to hepatocellular carcinoma. Dig Liver Dis. 2013 Sep;45(9):712-23. doi: 10.1016/j.dld.2013.01.012. Epub 2013 Feb 23. PMID 23769756